CLINICAL TRIAL: NCT04265612
Title: Effect of the Negative Pressure Therapy Dressing Compared With the Hydrogel Dressing on Surgical Wound Infection in Cardiac Surgery.
Brief Title: Effect of the Negative Pressure Therapy Dressing Compared With Hydrogel Dressing.
Acronym: PICO/2019
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds preventing further payment of the trial insurance
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PICO/2019
Record Dates: First submitted 2019-11-05; First posted 2020-02-11 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2021-02

CONDITIONS: Wound Infection, Surgical
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator
Masking Description: External evaluator: care provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure dressing (Experimental): Pico®" negative pressure dressing that will be placed in the operating room in both sternal wound and saphenectomy. This dressing will remain in place for 7 days without getting up, unless it has become saturated, in which case, only the dressing will be changed.
  Interventions: Procedure: Pico®" negative pressure dressing
- Aquacel hydrogel dressing (Active Comparator): Aquacel Surgical®" hydrogel dressing that will be placed in the operating room in both sternal wound and saphenectomy. This dressing will remain in place for 7 days without getting up, unless it has become saturated, in which case, only the dressing will be changed.
  Interventions: Procedure: Aquacel Surgical®" hydrogel dressing

INTERVENTIONS:
Procedure: Pico®" negative pressure dressing — Pico®" negative pressure dressing that will be placed in the operating room in both sternal wound and saphenectomy.The dressing will remain on for 7 days without waking up, unless it is saturated, in which case only the dressing will be changed
  Arms: Negative Pressure dressing
Procedure: Aquacel Surgical®" hydrogel dressing — Aquacel Surgical®" hydrogel dressing that will be placed in the operating room in both sternal wound and saphenectomy. This dressing will remain in place for 7 days without getting up, unless it has become saturated, in which case, only the dressing will be changed.
  Arms: Aquacel hydrogel dressing

SUMMARY:
The objective of the study is to measure the efficacy of the use of single-use portable negative pressure therapy (PICO ®) in the prevention of surgical wound infections (SSI) from cardiac surgery under extracorporeal circulation compared to single-use hydrocolloid dressings "Aquacel Surgical".

DETAILED DESCRIPTION:
Negative pressure therapy is a type of physical therapy for wound healing that is based on the application of a negative pressure (void) in the wound bed.

Negative pressure therapy is based on the application of a subatmospheric pressure in the wound bed to trigger a whole series of mechanisms, and that to a greater or lesser degree, and in a synergistic manner, act by creating or improving the conditions for the healing process to develop (negative pressure therapy).

All these mechanisms act by diminishing the possibility of creating an appropriate medium for the growth of pathogenic germs.

Today, negative pressure therapy is also used to create ideal conditions in surgical wounds to prevent or reduce the risk of local complications, is what we call incisional negative pressure therapy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective or emergency cardiac surgery with extracorporeal circulation heart surgery who will have a median sternotomy.
* Who signs Informed Consent after agreeing to participate in the microbiological study.

Exclusion Criteria:

* Patients undergoing emergency cardiac surgery that does not time to randomization and/or coding.
* Patients with immunocompromised haematological diseases.
* Patients who are allergic or present some hypersensitivity to the dressing or excipient.
* Patients who are participating in another experimental study.
* Patients who, due to their fragility or comorbidity, the surgeon considers that they should not undergo randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Incidence of infection of the sternal surgical wound. | 1-3 months
  The state of the surgical wound will be assessed and recorded on the wound care data collection sheet. Note whether the wound looks good or not and whether there are any complications: exudate, appearance of the wound, necrosis of the wound edges, redness, maceration of the wound or wound dehiscence.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez Sanz, PhD, Study Director — Hospital Universitario de Canarias; Pilar Garrido Martín, PhD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Pilar Garrido Martín, Santa Cruz de Tenerife, Spain